CLINICAL TRIAL: NCT02205177
Title: Expanding Access to Therapy for Childhood Anxiety Disorders Via Smart Phones - PILOT
Brief Title: Youth Mayo Clinic Anxiety Coach Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stephen Whiteside (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor-Investigator, Stephen Whiteside, Associate Professor of Psychology, Mayo Clinic
Organization: Mayo Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 13-000288 - PILOT; R34MH100468 (NIH)
Record Dates: First submitted 2014-07-29; First posted 2014-07-31 (Estimated); Results first posted 2019-08-05 (Actual); Last update posted 2019-08-05 (Actual); Status verified 2019-08

CONDITIONS: Anxiety
Keywords: Anxiety; Social Anxiety; Social Phobia; Separation Anxiety; Generalized Anxiety; GAD; Phobia; Panic; Agoraphobia; Obsessive Compulsive Disorder; OCD; Child; Adolescent; Smartphone; Teen; Youth
MeSH Terms: conditions — Anxiety Disorders; Phobia, Social; Anxiety, Separation; Generalized Anxiety Disorder; Phobic Disorders; Agoraphobia; Obsessive-Compulsive Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Face-to-Face w/ Anxiety Coach (FTF-AC) (Active Comparator): In this condition therapists will provide 6 to 12 50-minute, face-to-face therapy sessions using Anxiety Coach. The sessions are expected to initially occur weekly and be within the office although the therapist can leave the office to conduct exposure. The therapist is expected to utilize Anxiety Coach within the session, encourage the patient to use the application to complete homework, and review progress in-session via the web-based portal.
  Interventions: Device: Mayo Clinic Anxiety Coach
- Minimal Contact w/ Anxiety Coach (MC-AC) (Experimental): In this condition the therapist will meet with the patient and primary care giver for an initial 50-minute, face-to-face session to provide a tutorial on the use of Anxiety Coach. The therapist is expected to review the patient's progress via the web-based portal and communicate with the patient electronically at least once per week for a total of at least 6 and up to 12 weeks of intervention. Therapists will be allowed 2 additional face-to-face sessions if necessary and still remain in protocol.
  Interventions: Device: Mayo Clinic Anxiety Coach

INTERVENTIONS:
Device: Mayo Clinic Anxiety Coach — Mayo Clinic Anxiety Coach is a smartphone application based on cognitive-behavioral treatment for anxiety disorders (i.e., exposure-based therapy) that can be used as 1) a stand-alone treatment requiring minimal provider contact, and 2) an augmentation of face-to-face treatment that increases clinician fidelity and patient adherence to evidence-based treatment. The design of Anxiety Coach is based on evidence and theory suggesting that information and communication technologies (ICTs) are well-suited for encouraging behavior change through 1) scheduled reminders to engage in therapeutic exercises, 2) point of performance support, 3) individually tailored information, 4) real-time symptom assessment, and 5) readily accessible asynchronous communication.

SUMMARY:
This research study aims to test the feasibility and effectiveness of using the Mayo Clinic Anxiety Coach smartphone app as an addition to traditional therapy for the treatment of anxiety disorders in youth, particularly those youth who may have limited access to mental health treatment in the traditional clinical setting.

DETAILED DESCRIPTION:
This research study aims to test the feasibility and effectiveness of using the Mayo Clinic Anxiety Coach smartphone app as an addition to traditional therapy for the treatment of anxiety disorders in youth, particularly those youth who may have limited access to mental health treatment in the traditional clinical setting. Therapist will provide CBT to patients with infrequent face-to-face contact and then will examine the acceptability, ease of use and need for contact.

ELIGIBILITY:
Inclusion Criteria:

1. Age 7 to 17
2. Primary diagnosis of:

   1. social phobia,
   2. separation anxiety disorder,
   3. panic disorder with and without agoraphobia,
   4. specific phobia, or
   5. obsessive compulsive disorder
3. A parent or other primary care giver available to participate with the child in all assessment and treatment activities
4. Estimated average intelligence
5. English speaking

Exclusion Criteria:

1. History of and/or current diagnosis of:

   1. psychosis,
   2. autism,
   3. bipolar disorder,
   4. mental retardation,
   5. oppositional defiant disorder,
   6. PTSD,
   7. selective mutism, or
   8. major depressive disorder
2. Current suicidality or recent suicidal behavior
3. Parent to be involved in study who is unable to adequately participate due to intellectual or psychiatric difficulties
4. Starting or changing the dosage of a psychiatric medication in the last two months

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2016-01-15 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Whiteside, PhD, LP, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Face-to-Face w/ Anxiety Coach (FTF-AC): In this condition therapists will provide 6 to 12 50-minute, face-to-face therapy sessions using Anxiety Coach. The sessions are expected to initially occur weekly and be within the office although the therapist can leave the office to conduct exposure. The therapist is expected to utilize Anxiety Coach within the session, encourage the patient to use the application to complete homework, & review progress in-session via the web-based portal.
  Mayo Clinic Anxiety Coach is a smartphone application based on cognitive-behavioral treatment for anxiety disorders (i.e., exposure-based therapy) that can be used as 1) a stand-alone treatment requiring minimal provider contact, and 2) an augmentation of face-to-face treatment that increases clinician fidelity & patient adherence to evidence-based treatment. The design of Anxiety Coach is based on evidence & theory suggesting that information and communication technologies (ICTs) are well-suited for encouraging
- Minimal Contact w/ Anxiety Coach (MC-AC): In this condition the therapist will meet with the patient and primary care giver for an initial 50-minute, face-to-face session to provide a tutorial on the use of Anxiety Coach. The therapist is expected to review the patient's progress via the web-based portal and communicate with the patient electronically at least once per week for a total of at least 6 & up to 12 weeks of intervention. Therapists will be allowed 2 additional face-to-face sessions if necessary and still remain in protocol.
  Mayo Clinic Anxiety Coach: Mayo Clinic Anxiety Coach is a smartphone application based on cognitive-behavioral treatment for anxiety disorders (i.e., exposure-based therapy) that can be used as 1) a stand-alone treatment requiring minimal provider contact, and 2) an augmentation of face-to-face treatment that increases clinician fidelity and patient adherence to evidence-based treatment. The design of Anxiety Coach is based on evidence and theory suggesting that information and communicatio
Period: Overall Study
Arm/Group | Face-to-Face w/ Anxiety Coach (FTF-AC) | Minimal Contact w/ Anxiety Coach (MC-AC)
Started | 8 | 2
Completed | 6 | 2
Not Completed | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Face-to-Face w/ Anxiety Coach (FTF-AC): Therapists will provide 6 to 12 50-minute, face-to-face therapy sessions using Anxiety Coach. The sessions occur weekly & within the office. Therapists will use Anxiety Coach at each session, encouraging patients to use the application to complete homework, & review progress in-session via the web-based portal.
  Mayo Clinic Anxiety Coach, a smartphone application based on cognitive-behavioral treatment for anxiety disorders can be used as a stand-alone treatment using minimal provider contact & an augmentation of face-to-face treatment that increases clinician fidelity & patient adherence to evidence-based treatment. Anxiety Coach's design is based on evidence & theory suggesting that information & communication technologies (ICTs) are well-suited for encouraging behavior change through scheduled reminders to engage in therapeutic exercises; point of performance support; individually tailored information; real-time symptom assessment & readily accessible asynchronous communication.
- Minimal Contact w/ Anxiety Coach (MC-AC): Therapist's will meet with the patient & parent for an initial 50-minute, face-to-face session to give a tutorial on using Anxiety Coach. The therapist will review the patient's progress via the web-based portal & communicate with patients electronically weekly for a total of 6 to 12 weeks of intervention.
  Mayo Clinic Anxiety Coach, a smartphone application based on cognitive-behavioral treatment for anxiety disorders can be used as a stand-alone treatment using minimal provider contact & an augmentation of face-to-face treatment that increases clinician fidelity & patient adherence to evidence-based treatment. Anxiety Coach's design is based on evidence & theory suggesting that information & communication technologies (ICTs) are well-suited for encouraging behavior change through scheduled reminders to engage in therapeutic exercises; point of performance support; individually tailored information; real-time symptom assessment & readily accessible asynchronous communication.
- Total: Total of all reporting groups
Arm/Group | Face-to-Face w/ Anxiety Coach (FTF-AC) | Minimal Contact w/ Anxiety Coach (MC-AC) | Total
Number analyzed (Participants) | 8 | 2 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 8 | 2 | 10
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 7
  Male | 3 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 8 | 2 | 10
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Pediatric Anxiety Rating Scale (PARS) at Treatment Completion
Description: The Pediatric Anxiety Rating Scale (PARS) is an interview-based tool used to assess for the presence and severity of anxiety symptoms in children and adolescents utilizing parental and youth input to guide clinician ratings. The PARS has 5 questions. Four of those questions has a scale ranging from none (1) to extreme (5). The other question has a rating of 1-5. The total score ranges from 0 - 25, with 25 being the worst.
Time Frame: Within 5 working days of Treatment Completion
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Face-to-Face w/ Anxiety Coach (FTF-AC) | Minimal Contact w/ Anxiety Coach (MC-AC)
Number analyzed (Participants) | 8 | 2
score on a scale | 11 (3.1) | -1 (.7)

2. Secondary Outcome: Number of Participants Who Completed the Subject Safety and Treatment Adherence Interview
Description: The number of patients that completed the summary of the qualitative interview will be used to enhance Anxiety Coach
Time Frame: Within 5 working days of Treatment Completion
Population: No families from minimal contact responded to interview request. three of the families from the Face to Face condition did not respond to invitation to interview.
Measure: Count of Participants; unit: Participants
Arm/Group | Face-to-Face w/ Anxiety Coach (FTF-AC) | Minimal Contact w/ Anxiety Coach (MC-AC)
Number analyzed (Participants) | 5 | 0
Participants | 5 | 0

ADVERSE EVENTS:
Time Frame: 11 months
Arm/Group | Face-to-Face w/ Anxiety Coach (FTF-AC) | Minimal Contact w/ Anxiety Coach (MC-AC)
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/2
Other Adverse Events (participants affected / at risk) | 0/8 | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-07-01): https://cdn.clinicaltrials.gov/large-docs/77/NCT02205177/Prot_001.pdf
  • Statistical Analysis Plan (2019-07-01): https://cdn.clinicaltrials.gov/large-docs/77/NCT02205177/SAP_002.pdf